CLINICAL TRIAL: NCT00240214
Title: An Open Label Post Marketing Surveillance Assessment to Evaluate the Effectiveness and Safety of Rapamune in Patients After Kidney Transplantation Receiving a Rapamune Containing Regime
Brief Title: Study Evaluating Rapamune in Patients After Kidney Transplantation
Status: Terminated | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Other Study IDs: 0468E-100875
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2008-03-14 (Estimated); Status verified 2008-03

CONDITIONS: Renal Transplantation
Keywords: Kidney transplants
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: sirolimus
  Interventions: Drug: sirolimus

INTERVENTIONS:
Drug: sirolimus — Tablet, dosage is determined by trough level

SUMMARY:
The purpose of this study is to obtain data on the effectiveness and safety of Rapamune under everyday conditions

ELIGIBILITY:
Inclusion Criteria:

* Patients having received a renal allograft from a cadaveric or living donor with low or moderate risk of developing acute rejection episodes.

Exclusion Criteria:

* Contraindications according to Summary of the Product Characteristics (SmPC).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2001-04; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Germany, medinfoDEU@wyeth.com
Locations (1):
- Multiple Cities, Germany